CLINICAL TRIAL: NCT01159496
Title: A Randomized Investigator And Subject-Blind, Sponsor Open, Placebo Controlled Phase 1 Study To Characterize The Safety, Tolerability, And Pharmacokinetics Of Ascending Multiple Doses Of PF-05212377 (SAM-760) Administered Orally To Healthy Young And Elderly Subjects
Brief Title: Multiple Ascending Dose Study To Assess Safety, Tolerability And Pharmacokinetics Of PF-05212377 (SAM-760)
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: B2081003
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
MeSH Terms: interventions — SAM-760

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: PF-05212377 (SAM-760)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05212377 (SAM-760) — Oral capsule, once daily for 14 days 1.5 mg, 5 mg, 15 mg, 30 mg and 50 mg
  Other Names: SAM-760
  Arms: Active
Drug: Placebo — Oral capsule, once daily for 14 days
  Arms: Placebo

SUMMARY:
This is a multiple ascending dose study to assess the safety, tolerability and pharmacokinetics of PF-05212377 (SAM-760) administered orally once a day for 14 days to healthy young adults and healthy elderly subjects. The study will be conducted under double-blind conditions (neither the investigator nor the subject will know if he/she has received PF-05212377 or a placebo). The Sponsor will know if the subject has received active treatment or a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for young healthy population: Healthy male and/or female subjects of non-child bearing potential (WONCBP) between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified at screening by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12-lead ECG, neurological examination and clinical laboratory tests.)
* Inclusion Criteria for elderly population: Healthy male and/or female subjects of non-child bearing potential between the ages of 65 and 85 years, inclusive. Subjects must be in reasonably good health as determined by the investigator based on a detailed medical history, full physical examination (including blood pressure and pulse rate measurement), 12-lead ECG and clinical laboratory tests. Subjects with mild, chronic, stable disease (eg, controlled hypertension, non-insulin dependent diabetes, osteoarthritis) may be enrolled if deemed medically prudent by the investigator.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* A score of greater than or equal to 20 on the Beck Depression Inventory and/or a response of 1, 2, or 3 to the question related to suicide.
* History of seizure disorder and/or severe head trauma (other than a single childhood febrile seizure).
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, dermatologic, muscular or allergic disease or disorder (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the study treatment.
* Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before study Day 1.
* History of drug abuse within 1 year before study Day 1 or a positive urine drug screen.
* Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements.
* Consumption of more than 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Subjects who smoke more than 10 cigarettes per day.
* Pregnant or nursing females; females of childbearing potential.
* Males who are unwilling to abstain from sexual intercourse or use a condom with all child-bearing potential women for the duration of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse events (spontaneous and solicited). | 0-24days
Change from baseline in vital signs. | 0-24 days
Change from baseline in triplicate ECGs. | 0-24 days
Clinical safety laboratory endpoints, including a complete blood count, reticulocytes and a full chemistry panel, including electrolytes, hepatic transaminases, and urinalysis, with microscopic analysis if dipstick analysis is positive. | 0-24 days
Physical examinations and neurological examinations | 0-24 days

SECONDARY OUTCOMES:
Pharmacokinetics in young adults (Plasma concentration of PF-05212377 over time (eg, AUC, Cmax, Tmax, t1/2). | 0-21 days
Pharmacokinetics in elderly subjects (Plasma concentration of PF-05212377 over time (eg, AUC, Cmax, Tmax, t1/2). | 0-21 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Rueil-Malmaison, France

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2081003&StudyName=Multiple%20Ascending%20Dose%20Study%20To%20Assess%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20PF-05212377%20%28SAM-760%29